CLINICAL TRIAL: NCT03944122
Title: Comparing the Efficacy of Continuous and Pulsed Ultrasound Treatments in Patients With Lateral Epicondylitis : a Double Blind, Randomized and Placebo-controlled Study
Brief Title: Comparing the Efficacy of Continuous and Pulsed Ultrasound Treatments in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Onur Armağan, Onur Armagan, medical doctor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FTR
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis, therapeutical ultrasound
MeSH Terms: conditions — Tennis Elbow | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: the patients and the physician was blind to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- continuous ultrasound (Experimental): continuous ultrasound were applied to the patients
  Interventions: Device: ultrasound
- pulsed ultrasound (Experimental): pulsed ultrasound were applied to the patients
  Interventions: Device: ultrasound
- placebo (Experimental): placebo (sham) ultrasound were applied to the patients
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — therapeutical ultrasound were applied to the patients

SUMMARY:
Objectives: The purpose of this study was to investigate the efficacy of continuous and pulsed ultrasound treatments in lateral epicondylitis and to compare the efficacy of these two treatments against each other and placebo.

Patients and Methods: Fifty one patients diagnosed with lateral epicondylitis were included to the study. Patients were randomised to continuous ultrasound, pulsed ultrasound and placebo groups by using closed envelop method. First group received continuous ultrasound treatment. Second group received pulsed ultrasound treatment in proportion as. Third group received of placebo treatment. Resting and moving pain levels of the patients were evaluated by using visual analog scale. Muscle strength was evaluated by using dynamometer. For functional evaluation Duruoz's hand index and Patient-Rated Tennis Elbow Evaluation (PRTEE) scales were used. Evaluations were made at baseline, at the end of the therapy, and one month after the therapy. In addition, at baseline and at the end of the therapy, the thickness of the common extensor tendon was measured by using ultrasonic imaging (USG).

DETAILED DESCRIPTION:
The purpose of this study was to investigate the efficacy of continuous and pulsed ultrasound treatments in lateral epicondylitis and to compare the efficacy of these two treatments against each other and placebo.

Fifty one patients (33 women, 18 men) diagnosed with lateral epicondylitis were included to the study. Patients were randomised to continuous ultrasound (n=17), pulsed ultrasound (n=17) and placebo (n=17) groups by using closed envelop method. First group received 10 sessions of 1 W/cm2 and 1,5 MHz continuous ultrasound treatment. Second group received 10 sessions of 1 W/cm2 and 1,5 MHz pulsed ultrasound treatment in proportion as 1:4. Third group received 10 sessions of placebo treatment with the same device seemed to be working but without delivering any output. Resting and moving pain levels of the patients were evaluated by using visual analog scale. Muscle strength was evaluated by using dynamometer. For functional evaluation Duruoz's hand index and Patient-Rated Tennis Elbow Evaluation (PRTEE) scales were used. Evaluations were made at baseline, at the end of the therapy, and one month after the therapy. In addition, at baseline and at the end of the therapy, the thickness of the common extensor tendon was measured by using ultrasonic imaging (USG).

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-70 years
* pain on the lateral side of the elbow for less than six months
* tenderness over the lateral epicondyle
* pain during extension of wrist and fingers

Exclusion Criteria:

* upper extremity and neck disorders
* other elbow pathologies
* presence of tendon rupture
* usage of non-steroidal anti inflammatory drugs
* joint limitations due to a previous radius/ulna fracture
* previous elbow surgery
* osteoporosis, malignancy, hemophilia, neurologic deficit(s) in the ipsilateral upper limb
* cognitive disfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-05-05 (Actual); Primary Completion 2015-05-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
measuring the thickness of common extensor tendon by ultrasound imaging. | 2nd week
  the thickness of common extensor tendon by ultrasound imaging was measured at the beginning and at the end of the study

SECONDARY OUTCOMES:
Visual Analog Scale | 6th week
Duruoz's hand index | 6th week
Patient-Rated Tennis Elbow Evaluation (PRTEE) scales | 6th week

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakılan, Study Director — Eskisehir City Hospital